CLINICAL TRIAL: NCT02619240
Title: Application of GeneXpert on Bronchoscopic Samples in the Clinical Management of Patients Suspicious of TB
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, To Kin Wang, Doctor, Chinese University of Hong Kong
Other Study IDs: CREC 2014.556
Record Dates: First submitted 2015-11-23; First posted 2015-12-02 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bronchoscopic alveolar lavage

GROUPS / COHORTS (1):
- patients suspected of TB: patients suspected of TB requiring to undergo bronchoscopy as part of the investigation
  Interventions: Procedure: bronchoscopy

INTERVENTIONS:
Procedure: bronchoscopy — performance of bronchoscopy with BAL

SUMMARY:
This is a case control observational study using Bronchial-alveolar lavage (BAL) as specimen for GeneXpert, a real time polymerase chain reaction (PCR) test for detection of tuberculosis (TB). Patients suspicious of TB, who require bronchoscopy as part of the investigation procedures, will be recruited for this study over a period of 18 months. Clinical likelihood of TB will be systematically scored according to various clinical parameters. This will determine the pre-test probability. Clinician will decide if anti-TB treatment is to be started and patients will be followed up for a minimal of 18 months. Sensitivity, specificity, positive, negative predictive values and the respective likelihood ratio will be calculated accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years old suspected of TB clinically.
2. Patients suspected of TB but both smear microscopy and TB PCR of sputum are negative or sputum cannot be produced.
3. BAL samples obtained following standard investigation procedure
4. CXR or CT imaging available.

Exclusion Criteria:

1. Bronchoscopy is not planned as a necessary procedure for investigation.
2. Diagnosis of active TB has been made by other means.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult patients with abnormal chest imaging suspected of TB as a differential diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-04-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
The number of true positive BAL PCR using GeneXpert on BAL for rapid diagnosis of TB in few hours compare to the conventional TB PCR which usually take up few days to perform | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kin Wang To, MBChB, Principal Investigator — Honoary clinical assistant professor
Locations (1):
- Department of Medicine and Therapeutics, Prince of Wales Hospital, CUHK, Shatin, Hong Kong